CLINICAL TRIAL: NCT05137938
Title: Safety and Clinical Effects of Intranasal Ketamine in Ultra-REsistant Depression (SURE-ECT Non Responders). Pilot Study
Brief Title: Intranasal Ketamine in Ultra-REsistant Depression (SURE-ECT Non Responders)
Acronym: SURE-ECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 095-2019
Record Dates: First submitted 2021-11-02; First posted 2021-11-30 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Depression
Keywords: Convulsive therapy; Open-label trial; Pilot study; Treatment-resistant depression (TRD); Ketamine; Intranasal drug delivery (IN); N-methyl-d-aspartate (NMDA); Receptor antagonist; Transcranial magnetic stimulation (TMS); Electromyography (EMG); Electroencephalography (EEG); Intracortical facilitation (ICF); Short-interval cortical inhibition (SICI); Electroconvulsive Therapy (ECT)
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: Open label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intranasal Ketamine (IN) (Experimental): Ketamine will be administered intranasally (IN) using an atomizer (MAD300 by Teleflex, North Carolina, USA).
  Interventions: Drug: Intranasal Ketamine (IN)

INTERVENTIONS:
Drug: Intranasal Ketamine (IN) — A sterile form of ketamine will be administered intranasally twice weekly for four weeks. Dosing schedule will be determined based on patient's weight using a specialized formula. Patients will be started at the lowest dose during the first treatment session. Dose will be titrated further to therapeutic dose in the following sessions. The dose will be adjusted if patients do not tolerate full therapeutic doses. After receiving the second treatment of each week, participants will be seen by a study physician to determine dosing for the following week. Patients will be monitored by trained personnel for the full duration of the 2 hour supervision period. Vital signs and physical symptoms will be monitored consistently and measurements taken every 30 minutes. Appropriate medications will be provided to manage treatment-related side effects and any adverse events. Labetalol will be used in the management of treatment-related transient hypertension as needed.

SUMMARY:
Despite the known efficacy of pharmacotherapy (i.e. antidepressants) and psychotherapeutic interventions in treating depressive disorders, research evidence suggests that 20% to 40% of patients with major depressive disorder (MDD) do not respond adequately to such treatments. These patients are diagnosed with Treatment-Resistant Depression (TRD), and are sometimes treated with convulsive therapy. However, about 10-30% of TRD patients do not respond to convulsive therapy, and are thus diagnosed with Ultra-Resistant Depression (URD). Using an open label pilot study involving subjects, this trial aims to assess the safety, tolerability, and clinical effects of intranasal ketamine (IN) treatment in patients who do not respond to convulsive therapy. Intranasal ketamine (IN) treatment approach has shown promising therapeutic outcomes for patients with TRD, but has not yet been studied on patients with URD.

DETAILED DESCRIPTION:
Ketamine is a fast-acting anesthetic that can have stimulant effects when taken at low doses. It acts as a non-competitive high-affinity N-methyl-d-aspartate (NMDA) receptor antagonist that stimulates synaptic glutamate release and blocks extra-synaptic NMDA receptors. This mechanism of action mediates excitatory synaptic transmission through the central nervous system and therefore results in robust antidepressant effects. Administering intravenous (IV) ketamine to patients with TRD has shown to produce rapid antidepressant effects. Nevertheless, delivering IV ketamine to patients can be challenging since it requires specialized expertise and equipment. A promising alternative that preserves IV ketamine's rapid onset of therapeutic action while minimizing inconvenience and discomfort is intranasal drug delivery (IN). This current proof-of-concept clinical trial is an open label pilot study on patients with treatment-resistant unipolar depression who did not respond to, or did not tolerate, an acute course of convulsive therapy. Using a combination of Transcranial Magnetic Stimulation (TMS) neurophysiological tools with electromyography (EMG) and electroencephalography (EEG), this trial also aims to explore biomarkers of ketamine's antidepressant effect by examining ketamine's action on NMDA neurotransmission. Investigating the impact of ketamine on cortical excitation and inhibition could provide insight into the role of NMDA receptors in cortical physiology, and therefore determine potential predictors of clinical response for depression.

Objective 1: To test the safety and tolerability of IN ketamine in patients with URD who did not respond to/tolerate an acute course of convulsive therapy

Hypothesis 1: IN ketamine will be safe and well tolerated in patients with URD

Objective 2: To test the clinical effects of IN ketamine patients with URD who did not respond to/tolerate an acute course of convulsive therapy

Hypothesis 2: IN ketamine will result in improvement in depressive symptoms, suicidal ideation, and quality of life measures (compared to scores from baseline)

Objective 3: To investigate the impact of ketamine on cortical excitation via intracortical facilitation (ICF) and cortical inhibition via short-interval cortical inhibition (SICI) paradigms

Hypothesis 3: IN ketamine will result in neurophysiological changes as measured by TMS-EMG and EEG

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with a diagnosis of non-psychotic MDD as confirmed by the Mini-International Neuropsychiatric Interview (MINI)
2. Individuals meeting criteria for Ultra Resistant Major Depressive Disorder (URD) in current episode

   URD is defined as:
   1. those who received at least eight convulsive therapy treatment sessions and did not respond, or
   2. those who were not able to tolerate convulsive therapy
3. Individuals scoring 14 and above on the Hamilton Rating Scale for Depression-24 Items (HRSD-24)
4. Individuals capable to provide consent who are receiving care as outpatients

Exclusion Criteria:

1. Individuals with history of substance use disorder (i.e. dependence or abuse) within the past month; and lifetime history of ketamine substance use disorder as confirmed by the MINI
2. Concomitant major unstable medical illness such as poorly controlled high blood pressure or patients diagnosed with enlarged prostate or reporting any other urinary related issues
3. Pregnancy or the intention to become pregnant and breastfeeding during the study as confirmed by self-report. Female participants of reproductive potential must be willing to use a medically acceptable method of birth control which include highly effective (e.g. approved hormonal contraceptives, intrauterine device, tubal ligation) or double barrier (e.g. male condom with diaphragm, male condom with cervical cap) methods of contraception or abstinence if that is the usual and preferred lifestyle of the participant
4. Presence of cardiac decompensation/heart failure v)
5. Diagnosis of any primary psychotic disorder, bipolar disorder, obsessive-compulsive disorder, or post-traumatic stress disorder (current) as confirmed by the MINI
6. Diagnosis of severe personality disorder as assessed during the initial consultation with a physician at the Temerty Centre prior to study entry
7. Any significant neurological disorder (e.g., a space occupying brain lesion, a history of stroke, a cerebral aneurysm, a seizure disorder, Parkinson's disease, Huntington's chorea, multiple sclerosis) as assessed through medical history review during the initial consultation with a physician at the Temerty Centre prior to study entry
8. Individuals presenting with a medical condition, a medication, or a laboratory abnormality that could cause a major depressive episode or significant cognitive impairment in the opinion of the investigator
9. Individuals requiring a benzodiazepine with a dose equivalent to lorazepam 2 mg/day or higher; being on any anticonvulsant(e.g. Lamotrigine) and/or opioid medication due to the potential of these medications to limit the efficacy of ketamine
10. Individuals unable to communicate in spoken and written English fluently enough to complete the required study assessments due to a language barrier or a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete clinical assessments)
11. Individuals with cognitive or physical impairment which may potentially interfere with IN ketamine administration and subject's ability to stay in the same place for a 2-hr monitoring supervision as assessed through medical history review during the initial consultation with a physician at the Temerty Centre prior to study entry
12. Any intracranial implant (e.g., aneurysm clips, shunts, cochlear implants) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed given that we will be using TMS-EMG/EEG
13. Those unable to secure escort to accompany them back home after ketamine sessions will also be excluded from this study
14. Any known allergy to the study medication or any component/ingredient of the ketamine preparation

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Change in symptom severity of depression as measured by the Hamilton Rating Scale for Depression - 24 | 2 months
  Hamilton Rating Scale for Depression (24-item version); This scale is used to quantify the severity of symptoms of depression Scale range: 0-76 (total score) Lower scores indicate lower severity of depressive symptoms (i.e., better outcome) Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)

SECONDARY OUTCOMES:
Change in symptom severity of Suicidal Ideation as measured by by the Scale of Suicide Ideation (SSI) | 2 months
  Scale for Suicide Ideation (SSI); This scale is used to assess the presence or absence of suicidal ideation and the degree of severity of suicidal ideas Scale range: 0-38 (total score) Lower scores indicate lower severity of suicidal ideation (i.e., better outcome) Higher scores indicate higher severity of suicidal ideation (i.e., worse outcome)
Safety and tolerability as assessed by changes in Blood Pressure (BP) | 1 month
  Assessed through monitoring of systolic and diastolic Blood Pressure (mmHg) on each treatment session before treatment and every 30 minutes within a 2-hour monitoring period.
Safety and tolerability as assessed by changes in Heart Rate (BPM) | 1 month
  Assessed through monitoring of Heart Rate (beats per minute) on each treatment session before treatment and every 30 minutes within a 2-hour monitoring period.
Safety and tolerability as assessed by changes in O2 Saturation | 1 month
  Assessed through monitoring of Oxygen saturation levels on each treatment session before treatment and every 30 minutes within a 2-hour monitoring period.
Safety and Tolerability of IN Ketamine as assessed by monitoring of adverse events | 2 months
  Assessed through monitoring of adverse events, cardiovascular adverse events and/or respiratory distress throughout the trial.
Impact of Ketamine on cortical excitation as measured by intracortical facilitation (ICF) | 1 months
  Assessed through administration of neurophysiological paradigms using Transcranial Magnetic Stimulation (TMS) paired with electromyography (EMG) and electroencephalography (EEG).
Impact of Ketamine on cortical inhibition as measured by short-interval cortical inhibition (SICI) | 1 month
  Assessed through administration of neurophysiological paradigms using Transcranial Magnetic Stimulation (TMS) paired with electromyography (EMG) and electroencephalography (EEG).

OTHER OUTCOMES:
Change in quality of life measures as assessed by the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | 1 month
  World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) (12-item version); This scale is used to assess disability over six domains of functioning: cognition, mobility, self-care, getting along with others, participation in society, and life activities.
  Scale range: 12-60 (total score) Lower scores indicate lower disability or loss of function (i.e., better outcome) Higher scores indicate higher disability or loss of function (i.e., worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Yuliya Knyahnytska, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Knyahnytska Y, Zomorrodi R, Kaster T, Voineskos D, Trevizol A, Blumberger D. The Safety, Clinical, and Neurophysiological Effects of Intranasal Ketamine in Patients Who Do Not Respond to Electroconvulsive Therapy: Protocol for a Pilot, Open-Label Clinical Trial. JMIR Res Protoc. 2022 Jan 17;11(1):e30163. doi: 10.2196/30163. PMID 34882570